CLINICAL TRIAL: NCT07230054
Title: Clinicopathological Features and Treatment Strategies for Gastric Epithelial Neoplasm of Fundic-gland Mucosa Lineage: A Multicenter Retrospective Study
Brief Title: Clinicopathological Features and Treatment Strategies for Gastric Epithelial Neoplasm of Fundic-gland Mucosa Lineage
Status: Completed | Type: Observational
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: NFEC-2024-644
Record Dates: First submitted 2025-07-22; First posted 2025-11-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Gastric Epithelial Neoplasm of Fundic-gland Mucosa
Keywords: Gastric epithelial neoplasm of fundic-gland mucosa lineage; oxyntic gland adenoma; gastric adenocarcinoma of fundic-gland type; gastric adenocarcinoma of fundic-gland mucosa type

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- oxyntic gland adenoma: Cases were diagnosed as OGA according to the histological and immunohistochemical diagnostic criteria for low-grade dysplasia and differentiated gastric cancer established in previous studies.
- gastric adenocarcinoma of fundic-gland type: Cases were diagnosed as GA-FG according to the histological and immunohistochemical diagnostic criteria for low-grade dysplasia and differentiated gastric cancer established in previous studies.
- gastric adenocarcinoma of fundic-gland mucosa type: Cases were diagnosed as GA-FGM according to the histological and immunohistochemical diagnostic criteria for low-grade dysplasia and differentiated gastric cancer established in previous studies.

SUMMARY:
Gastric epithelial neoplasm of fundic-gland mucosa lineage (GEN-FGML) is a rare pathological type of gastric cancer characterized by unique endoscopic features, including specific morphology, color, and changes in the surface and vascular patterns of the lesion. Histologically, GEN-FGML is an epithelial neoplasm exhibiting gastric fundic gland differentiation. Based on cellular differentiation and submucosal invasion, it can be classified into three subtypes:

1. Oxyntic gland adenoma (OGA);
2. Gastric adenocarcinoma of fundic-gland type (GA-FG);
3. Gastric adenocarcinoma of fundic-gland mucosa type (GA-FGM). GA-FGM can be further subdivided into three subtypes: Type 1 (regular exposed pattern), Type 2 (disordered exposed pattern), and Type 3 (disordered non-exposed pattern).

Some studies have analyzed the clinicopathological characteristics, endoscopic features, molecular biological characteristics, treatment strategies, and prognosis of the different GEN-FGML subtypes. Generally, OGA and GA-FG present as low-grade epithelial neoplasms with a favorable prognosis, whereas GA-FGM exhibits higher rates of lymphovascular invasion and behaves as a high-grade malignant tumor.However, due to the currently limited number of reported cases, there are no international guidelines or consensus regarding the selection of treatment strategies for GEN-FGML, curative resection evaluation, and prognosis.

In this study, the investigators aim to retrospectively collect data on GEN-FGML cases from multiple centers in China and compare the clinicopathological characteristics, molecular biological features, endoscopic characteristics, treatment strategies, and patient prognosis among the different GEN-FGML subtypes.

DETAILED DESCRIPTION:
1. Research Background

Gastric epithelial neoplasm of fundic-gland mucosa lineage (GEN-FGML) is a rare pathological type of gastric cancer characterized by unique endoscopic features, including specific morphology, color, and changes in the surface and vascular patterns of the lesion. In 2007, Tsukamoto et al. reported the first case of gastric adenocarcinoma with chief cell differentiation. In 2010, Ueyama et al. proposed gastric adenocarcinoma of fundic-gland type (GA-FG) as a novel variant of gastric adenocarcinoma. Subsequently, gastric adenocarcinoma of fundic-gland mucosa type (GA-FGM) was also reported; this subtype exhibits gastric foveolar epithelial differentiation in addition to fundic gland differentiation and demonstrates more aggressive behavior.Histologically, GEN-FGML is an epithelial neoplasm exhibiting gastric fundic gland differentiation. Based on cellular differentiation and submucosal invasion, it can be classified into three subtypes:

1. Oxyntic gland adenoma (OGA);
2. Gastric adenocarcinoma of fundic-gland type (GA-FG);
3. Gastric adenocarcinoma of fundic-gland mucosa type (GA-FGM). GA-FGM can be further subdivided into three subtypes: Type 1 (regular exposed pattern), Type 2 (disordered exposed pattern), and Type 3 (disordered non-exposed pattern).

Some studies have analyzed the clinicopathological characteristics, endoscopic features, molecular biological characteristics, treatment strategies, and prognosis of the different GEN-FGML subtypes. Generally, OGA and GA-FG present as low-grade epithelial neoplasms with a favorable prognosis, whereas GA-FGM exhibits higher rates of lymphovascular invasion and behaves as a high-grade malignant tumor.

However, due to the currently limited number of reported cases, there are no international guidelines or consensus regarding the selection of treatment strategies for GEN-FGML, curative resection evaluation, and prognosis. Furthermore, the majority of reported cases have been described by Japanese researchers, and data on the incidence, detection rate, treatment strategies, and clinical prognosis of GEN-FGML in other countries remain scarce.

Based on this, there is an urgent need for systematic research into the clinicopathological characteristics, endoscopic features, treatment strategies, and prognosis of GEN-FGML. This study aims to provide high-quality, evidence-based medical evidence to inform the development of standardized treatment strategies, curative evaluation, and prognostic assessment for GEN-FGML. Specifically, the investigators aim to retrospectively collect data on GEN-FGML cases from multiple centers in China and compare the clinicopathological characteristics, molecular biological features, endoscopic characteristics, treatment strategies, and patient prognosis among the different GEN-FGML subtypes.

2. Research Objectives

The objectives of this study are to:

1. Retrospectively collect cases and clinical data related to GEN-FGML from multiple centers across China.
2. Compare the clinicopathological characteristics, endoscopic features, molecular biological characteristics, clinical treatment modalities, and patient prognosis among the different subtypes of GEN-FGML.
3. Provide high-quality, evidence-based data to support the development of standardized treatment strategies, curative resection evaluation, and prognostic assessment for GEN-FGML.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who voluntarily provided written informed consent between August 1, 2010 and August 1, 2024
2. Age ≥18 years at diagnosis
3. Confirmed diagnosis of GEN-FGML

Exclusion Criteria:

* The clinicopathological data of the lesion(s) were missing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who confirmed diagnosis of GEN-FGML
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2010-08-01 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Comparison of Clinicopathological Characteristics Among Different Subtypes of GEN-FGML | From enrollment to the end of treatment at 2 years
  Data extracted from Electronic Medical Records (EMRs):
  Imaging Results (CT)
Comparison of Clinicopathological Characteristics Among Different Subtypes of GEN-FGML | From enrollment to the end of treatment at 2 years
  Endoscopic Findings(presence of atrophic gastritis, lesion location, lesion size, lesion color, gross morphology of the lesion, presence of lesion borders, presence of mucosal atrophy around the lesion, presence of dilated branching vessels, regularity of lesion color, regularity of the mucosal structure on the lesion surface, presence of granular changes in the lesion mucosa)
Comparison of Clinicopathological Characteristics Among Different Subtypes of GEN-FGML | From enrollment to the end of treatment at 2 years
  Histopathological Results[the type of GEN-FGML:OGA, GA-FG, GA-FGM. result of immunohistochemistry(positve or negative): MUC5AC, MUC6, MUC2, CD10, p53, H+K+-ATP，Ki-67]
Comparison of Therapeutic Approaches Among Different Subtypes of GEN-FGML | From enrollment to the end of treatment at 2 years
  Treatment Modalities(Endoscopic forceps removal, cold resection, snare electrosurgical resection, endoscopic mucosal resection, endoscopic submucosal dissection , surgical surgery）
Comparison of Prognosis Among Different Subtypes of GEN-FGML | From enrollment to the end of treatment at 2 years
  Surveillance（including Endoscopic Surveillance and Imaging Surveillance )

SECONDARY OUTCOMES:
Medical of GEN-FGML Patients. | From enrollment to the end of treatment at 2 years
  Data extracted from Electronic Medical Records (EMRs): Medical History（age、clinical symtoms such as acid reflux, heartburn, and abdominal pain)

CONTACTS AND LOCATIONS:
Locations (1):
- Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No